CLINICAL TRIAL: NCT02137408
Title: Docosahexaenoic Acid Supplementation of Women With Hypertension in Pregnancy to Improve Endothelial Health and Reduce the Risks of Preterm Delivery
Brief Title: Docosahexaenoic Acid Supplementation of Women With Hypertension in Pregnancy to Improve Endothelial Health
Acronym: DHA-2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at Institution
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-7329
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension in Pregnancy
Keywords: Chronic hypertension in pregnancy; Pre-term delivery; Preeclampsia; Endothelial Health; Docosahexaenoic acid (DHA)
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 200 mg docosahexaenoic acid (Active Comparator): Participants will be randomized to 200 mg of docosahexaenoic acid (DHA) administered PO daily (1-200mg capsule of DHA). This is a standard dose used in prenatal vitamins. Participants will be supplemented by mouth daily between 18-20 weeks gestation through 6 weeks post-partum.
  Interventions: Dietary Supplement: Docosahexaenoic acid 200 mg
- 1000 mg docosahexaenoic acid (Active Comparator): Participants will be randomized to 1000 mg of docosahexaenoic acid (DHA) administered PO daily (5- 200mg capsules of DHA). Participants will be supplemented daily PO between 18-20 weeks gestation through 6 weeks post-partum.
  Interventions: Drug: Docosahexaenoic acid 1000 mg

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid 200 mg — Participants will be randomized to 200 mg docosahexaenoic acid daily (1-200mg capsule) PO beginning at 18-20 weeks gestation through 6 weeks post-partum.
  Other Names: 200mg dietary DHA daily (Expecta, Mead Johnson) PO
  Arms: 200 mg docosahexaenoic acid
Drug: Docosahexaenoic acid 1000 mg — Participants will be randomized to 1000 mg (5-200mg capsules) docosahexaenoic acid PO daily beginning at 18-20 weeks gestation through 6 weeks post-partum.
  Other Names: Dietary DHA (Expecta, Mead Johnson) will be given PO with 5-200mg capsules
  Arms: 1000 mg docosahexaenoic acid

SUMMARY:
The Investigator would like to see if taking a DHA supplement at a dose recommended for heart health will improve brachial artery dilation (relaxation) and help blood pressure. As a second goal the Investigator would like to see if this supplement can delay preterm delivery by improving heart health. In this research study, the Investigator is asking pregnant women with chronic high blood pressure to take Expecta (DHA - Martek Biosciences, now known as DSM Nutritional Lipil) during the last half of their pregnancy until six weeks after they deliver their baby.

DETAILED DESCRIPTION:
The Investigator will be supplementing pregnant mothers with Expecta. This is an over the counter supplement often used by pregnant and nursing mothers and will be given to expectant mothers during the research study. This DHA supplement is available to anyone at most any store. The dose often used over the counter is 200mg, we are testing the heart recommended dose of 1000mg. Because the Investigator is using the heart health recommended dose and because there may be a health claim, the Investigator is doing the study using an FDA- food and drug administration IND. IND means investigational drug. This dose has recently been used safely and effectively in pregnancy both here in the United States and in Australia in hundreds of women. There are no risks to the fetus as the placenta prefers to transfer this important nutrient for fetal eye and brain development. The large studies done in pregnancy have followed their babies into school age and found no adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women coming for their 19-20 week ultrasound for fetal anatomy and that have been diagnosed with hypertension by their Obstetrician will be eligible for inclusion.

Exclusion Criteria:

* Exclusions to enrollment will include: women < 18 years old
* Bleeding disorders
* Lupus
* Autoimmune diseases
* The presence of infant congenital (trisomy 13,18, 21, urethral, gastrointestinal and cardiac defects)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Improve maternal endothelial health | Pregnant mothers 18-20 weeks gestation (Baseline) - Six weeks post partum
  To test this hypothesis, the Investigator will undertake a RCT of 90 women with hypertension (chronic or newly diagnosed) in the second trimester of pregnancy, who will be randomized to 1000mg DHA or standard supplement and followed through to delivery with serial measures of blood pressure and vascular constriction by the Doppler method.

SECONDARY OUTCOMES:
Improve immune homeostasis | Pregnant mothers 18-20 weeks gestation (Baseline) through 6 weeks post partum
  Measured by decreased maternal blood and cord blood concentrations of pro-inflammatory cytokines IL-6, I L-8, TNF a, and receptor sRAGE.

OTHER OUTCOMES:
Decrease the number of infants born <34 weeks | Pregnant mothers 18-20 weeks gestation (Baseline) through 6 weeks post partum
  In addition to the primary aims, we will examine evidence that DHA will prolong gestation

CONTACTS AND LOCATIONS:
Overall Officials: Christina J Valentine, MD, MS, RD, Principal Investigator — Cincinnati Children's Hosptial Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States